CLINICAL TRIAL: NCT00426855
Title: Weekly Bendamustine and Bortezomib Combination Therapy in Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma or B-CLL: A Single-Center Phase 2 Study
Brief Title: Bendamustine and Bortezomib Combination Therapy in Indolent Non-Hodgkin's Lymphoma(NHL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter Moosmann (Other)
Collaborators: Kantonsspital Aarau (Other)
Responsible Party: Sponsor-Investigator, Peter Moosmann, MD PhD, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZOHT-01/07
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Lymphoma, Non-Hodgkin, Low-Grade
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Bendamustine Hydrochloride; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine and Bortezomib (Experimental): Combination Chemotherapy of Bendamustine and Bortezomib as described in the intervention section
  Interventions: Drug: Bendamustine; Drug: Bortezomib

INTERVENTIONS:
Drug: Bendamustine — starting with 60 mg/m^ 2, IV, dose escalation, weekly d1,8,15 q5w
  Other Names: Ribomustin, SDX-105
Drug: Bortezomib — weekly 1.5mg/m^2, IV, d1,8,15,22 q5w
  Other Names: Velcade

SUMMARY:
The purpose of this study is to determine whether the combination of bendamustine and bortezomib in patients with indolent Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia is safe and tolerable.

DETAILED DESCRIPTION:
Bendamustin and bortezomib have been shown to be effective in the treatment of patients with indolent Non-Hodgkin's Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL). Both compounds appear not to be cross-resistant with prior therapy. Therefore, it is of interest to combine bendamustine and bortezomib in this patient population.

Preliminary results from patients with multiple myeloma showed that the combination of bendamustine and bortezomib is efficacious and well tolerated. However, there are so far no data on this combination in patients with NHL or CLL.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic recurrent or refractory indolent NHL or B-CLL
* Adequate organ and bone marrow function
* Karnofsky greater than 50%

Exclusion Criteria:

* Candidates for autologous stem cell transplantation
* Secondary high grade lymphoma
* Concurrent severe medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Moosmann, MD PhD, Principal Investigator — Cantonal Hospital of Aarau, Switzerland

REFERENCES:
- [Result] Moosmann P, Heizmann M, Kotrubczik N, Wernli M, Bargetzi M. Weekly treatment with a combination of bortezomib and bendamustine in relapsed or refractory indolent non-Hodgkin lymphoma. Leuk Lymphoma. 2010 Jan;51(1):149-52. doi: 10.3109/10428190903275602. No abstract available. PMID 19860608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve consecutive patients of a medical clinic were included in the trial.
Groups:
- Group 1: Bortezomib, Bendamustine, NHL, combination chemotherapy
Period: Overall Study
Arm/Group | Group 1
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Bortezomib, Bendamustin, combination chemotherapy in nhl
Arm/Group | Group 1
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Optimal Bendamustine Dosage for Further Studies
Time Frame: Three weeks after treatment termination
Measure: Number; unit: mg/m^2
Groups:
- Group 1: NHL treated with combination chemotherapy of bendamustin and bortezomib
Arm/Group | Group 1
Number analyzed (Participants) | 12
mg/m^2 | 60

ADVERSE EVENTS:
Groups:
- Group 1: NHL Patients treated with combination of bendamustine and bortezomib
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=12)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=12)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 6 (6)
Dehydration (Cardiac disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Fatigue (Psychiatric disorders) | 6 (6)
Neuropathy, motor (Nervous system disorders) | 1 (1)
Neuropathy, sensory (Nervous system disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemorrhage, gastrointestinal (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No